CLINICAL TRIAL: NCT06286592
Title: CBPR Intervention to Decrease Lung Cancer Stigma and Health Disparities (LUNGevity Lung Cancer Stigma Reduction)
Brief Title: LUNGevity: Lung Cancer Stigma Community Based Participatory Research
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Kristen E. Riley, Ph.D., Assistant Professor, Clinical Psychology Department, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Pro2023002053
Record Dates: First submitted 2023-12-07; First posted 2024-02-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
Keywords: community-based participatory research; community advisory board; stimga; cancer; smoking cessation
MeSH Terms: conditions — Lung Neoplasms; Neoplasms; Smoking Cessation

STUDY DESIGN:
Intervention Model Description: Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Then, in a Phase IB trial, we will use a MOST design to assign patients to promising intervention components, combining them and altering exposure time, measuring preliminary effects of possible components of interventions. Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Conditions 1, 2 & 3 (Experimental): Condition 1 = Brief Mindfulness Video Condition 2 = Forgiveness Video Condition 3 = ACT Video
  *Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Interventions: Behavioral: Ultra-brief mindfulness intervention video; Behavioral: Forgiveness video; Behavioral: ACT values video
- Conditions 1 & 2 (Experimental): Condition 1 = Brief Mindfulness Video Condition 2 = Forgiveness Video
  *Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Interventions: Behavioral: Ultra-brief mindfulness intervention video; Behavioral: Forgiveness video
- Condition 1 (Experimental): Condition 1 = Brief Mindfulness Video
  *Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Interventions: Behavioral: Ultra-brief mindfulness intervention video
- Conditions 1 & 3 (Experimental): Condition 1 = Brief Mindfulness Video Condition 3 = ACT Video
  *Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Interventions: Behavioral: Ultra-brief mindfulness intervention video; Behavioral: ACT values video
- Conditions 2 & 3 (Experimental): Condition 2 = Forgiveness Video Condition 3 = ACT Video
  *Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Interventions: Behavioral: Forgiveness video; Behavioral: ACT values video
- Condition 2 (Experimental): Condition 2 = Forgiveness Video
  *Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Interventions: Behavioral: Forgiveness video
- Condition 3 (Experimental): Condition 3 = ACT Video
  *Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Interventions: Behavioral: ACT values video
- No Intervention (No Intervention): Treatment as usual.

INTERVENTIONS:
Behavioral: Ultra-brief mindfulness intervention video — Details of the specific intervention will be selected in collaboration with the Community Advisory Board.
  Then, in a Phase IB trial, we will use a MOST design to assign patients to promising intervention components, combining them and altering exposure time, measuring preliminary effects of possible components of interventions. Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Arms: Condition 1; Conditions 1 & 2; Conditions 1 & 3; Conditions 1, 2 & 3
Behavioral: Forgiveness video — Details of the specific intervention will be selected in collaboration with the Community Advisory Board.
  Then, in a Phase IB trial, we will use a MOST design to assign patients to promising intervention components, combining them and altering exposure time, measuring preliminary effects of possible components of interventions. Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Arms: Condition 2; Conditions 1 & 2; Conditions 1, 2 & 3; Conditions 2 & 3
Behavioral: ACT values video — Details of the specific intervention will be selected in collaboration with the Community Advisory Board.
  Then, in a Phase IB trial, we will use a MOST design to assign patients to promising intervention components, combining them and altering exposure time, measuring preliminary effects of possible components of interventions. Details of the specific interventions will be selected in collaboration with the Community Advisory Board.
  Arms: Condition 3; Conditions 1 & 3; Conditions 1, 2 & 3; Conditions 2 & 3

SUMMARY:
Lung cancer survival rates are low for intersectional underserved groups. Lung cancer stigma and intersectional stigma related to minoritized group status leads to increased morbidity and mortality and health disparities. Mindfulness interventions have been shown to decrease stigma and the negative impacts of stigma, however, these interventions have never been tested to decrease lung cancer stigma specifically. In this study, the investigators will use Community Based Participatory Research framework and MOST methodology to build and optimize a brief virtual mindfulness intervention to decrease lung cancer stigma, through first building a diverse coalition of lung cancer patients on a participatory action council.

DETAILED DESCRIPTION:
Lung cancer is the deadliest form of cancer, with the five year survival rate being 18.6%. Survival rates are even lower for intersectional underserved groups. Stigma about having lung cancer is very common, with 95% of lung cancer patients reporting lung cancer stigma. Stigma leads to higher rates of depressive symptoms, lower disclosure of smoking, lower likelihood of engaging with smoking cessation services, and decreased likelihood of following through on treatment recommendations. Lung cancer stigma and intersectional stigma related to minoritized group status leads to increased morbidity and mortality and health disparities. Mindfulness interventions have been shown to decrease stigma and the negative impacts of stigma, however, these interventions have never been tested to decrease lung cancer stigma specifically.

In this study, the investigators propose an innovative Multiphase Optimization Strategy (MOST) methodology to build and optimize a brief virtual mindfulness intervention to decrease lung cancer stigma. Using an innovative approach that combines Community Based Participatory Research (CBPR) and MOST, the investigators will first build a diverse coalition of lung cancer patients on a participatory action council per CBPR best practice models, with community members as equal stakeholders and part of the research team at every stage of the project. This study aims to:

Test mindfulness intervention components for lung cancer stigma in lung cancer patients to improve lung cancer treatment outcomes (i.e., patient-provider communication, willingness to accept referral to tobacco cessation, and quit rates).

Assess preliminary efficacy of these interventions on lung cancer stigma among lung cancer patients by race, ethnicity and sexual/gender classification.

Explore reach, acceptability and satisfaction of a mindfulness intervention to address lung cancer stigma, with a focus reaching patients in underserved groups (Black, Latinx, LGBTQ+ individuals, and low SES) in order to decrease health disparities and extend the five year survival rate.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be patients 18 years of age or older with a history of tobacco use to qualify for study inclusion. At least a portion of the participants will also need to be current lung cancer patients. Participants must be able to read and understand English and have normal to corrected vision and hearing.
* For the Community Advisory Board (CAB), participants must have been diagnosed with lung cancer, be at least 18 years of age or older, and self-identify as being part of an underrepresented group identity.

Exclusion Criteria:

* Any potential participants who do not meet the above inclusion criteria will be excluded from the study.
* Patients who are under the age of 18 and who do not have a history of tobacco use will be excluded from participating in the study.
* Individuals who cannot read or understand English or who do not have normal to corrected vision and hearing will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Lung Cancer Stigma Inventory (LCSI) | 1 year
  Both perceived/felt stigma (negative appraisal and devaluation from others) and internalized/self (internalization of perceived stigma) stigma from having lunch cancer.
Tobacco use quit likelihood | 1 year
  If current smoker, assessing subjectively reported quit likelihood on a 0 (meaning not likely) to 10 (meaning extremely likely) scale.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen E Riley, PhD, Principal Investigator — Rutgers, The State University of New Jersey

IPD SHARING:
Plan to Share IPD: Yes
Participant age range and status collected during trial will be reported after deidentification.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication. No end date.
Access Criteria: Anyone who wishes to access the data.

REFERENCES:
- [Background] Collins LM, Kugler KC, Gwadz MV. Optimization of Multicomponent Behavioral and Biobehavioral Interventions for the Prevention and Treatment of HIV/AIDS. AIDS Behav. 2016 Jan;20 Suppl 1(0 1):S197-214. doi: 10.1007/s10461-015-1145-4. PMID 26238037
- [Background] Sanchez V, Sanchez-Youngman S, Dickson E, Burgess E, Haozous E, Trickett E, Baker E, Wallerstein N. CBPR Implementation Framework for Community-Academic Partnerships. Am J Community Psychol. 2021 Jun;67(3-4):284-296. doi: 10.1002/ajcp.12506. Epub 2021 Apr 6. PMID 33823072
- [Background] Riley KE, Ulrich MR, Hamann HA, Ostroff JS. Decreasing Smoking but Increasing Stigma? Anti-tobacco Campaigns, Public Health, and Cancer Care. AMA J Ethics. 2017 May 1;19(5):475-485. doi: 10.1001/journalofethics.2017.19.5.msoc1-1705. PMID 28553905
- [Background] Vrinten C, Gallagher A, Waller J, Marlow LAV. Cancer stigma and cancer screening attendance: a population based survey in England. BMC Cancer. 2019 Jun 11;19(1):566. doi: 10.1186/s12885-019-5787-x. PMID 31185949
- [Result] Hatzenbuehler ML, Phelan JC, Link BG. Stigma as a fundamental cause of population health inequalities. Am J Public Health. 2013 May;103(5):813-21. doi: 10.2105/AJPH.2012.301069. Epub 2013 Mar 14. PMID 23488505